CLINICAL TRIAL: NCT05032794
Title: Unrestricted Diet vs 1-day Low Residue Diet for Screening Colonoscopy
Brief Title: Unrestricted Diet for Screening Colonoscopy
Acronym: CriLiP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc Taulí Hospital Universitari (Other)
Responsible Party: Principal Investigator, Salvador Machlab, Gastroenterology Consultant, Parc Taulí Hospital Universitari
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2021/3009
Record Dates: First submitted 2021-07-15; First posted 2021-09-02 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Bowel Cleansing; Colonoscopy; Bowel Cancer
Keywords: bowel cleansing; Diet; Low residue diet
MeSH Terms: conditions — Intestinal Neoplasms | interventions — Bisacodyl

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unrestricted diet (Experimental): The participant is not instructed to follow any dietary recommendation before colonoscopy. But only the restriction and fasting required for sedation.
  Interventions: Other: Unrestricted diet before colonoscopy; Drug: Bisacodyl 5 MG
- One day low residue diet (Active Comparator): The participant is instructed to follow a low residue diet the day before the colonoscopy.
  It will be given a informative document and educated by a nurse.
  Interventions: Other: 1-day low residue diet; Drug: Bisacodyl 5 MG

INTERVENTIONS:
Other: Unrestricted diet before colonoscopy — Free diet, without restrictions
  Arms: Unrestricted diet
Other: 1-day low residue diet — To follow a diet low in residues / fiber. the day before the colonoscopy.
  Arms: One day low residue diet
Drug: Bisacodyl 5 MG — If the participant is at risk of inadequate bowel cleansing, defined by a score of Dik et al ≥ 2 it will be given Bisacodyl 5 milgrams bid for 3 days.

SUMMARY:
Colonoscopy is the technique of choice for the evaluation of the mucosa of the colon. To be able to do the procedure in optimal conditions, it needs to be clean. Therefore, it is necessary to carry out a preparation as safe and tolerable as possible. This preparation generally consists in a low residue diet the days before the colonoscopy and in the intake of a laxative solution. In previous studies, it has been shown that the low residue diet does not play a relevant role as it was considered before. Recent studies demonstrated that reducing the days of low residue diet does not worsen the cleansing and improves the patient experience. The results of this study are required for determining the role of diet restrictive diet in colon cleansing.

ELIGIBILITY:
Inclusion Criteria:

* Individuals on the early colorectal cancer detection program who agreed to undergo colonoscopy after positive results on the fecal immunochemical test (FIT)

Exclusion Criteria:

* Individuals in which colonoscopy, cleansing solution or bisacodyl are contraindicated
* Subjects that are considered to have a linguistic barrier or to be unable to understand the instructions and / or give informed consent.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Adequate bowel cleansing | During colonoscopy (At the withdrawal phase)
  Bowel cleansing as a rating using the Boston Bowel Preparation Scale above 1 in each segment . This score ranges fron 0 to 3 in each one of the three segments. Zero is the worst outcome and 3 is the best cleansing

SECONDARY OUTCOMES:
Diet tolerability as assessed by a likert scale | The day of the colonoscopy just before beginning
  Tolerance to the diet assigned to the participant measured with a likert scale from 0 to 5, 0 the worst ad 5 the best.
Preparation tolerability as assessed by a likert scale and Hatoum et al. survey | The day of the colonoscopy just before beginning
  Tolerance to the cleansing solution used for bowel cleansing measured with a likert scale from 0 to 5, 0 the worst ad 5 the best.
  Hatoum et al is a validated survey designed for assessing bowel preparation tolerability DOI 10.1007/s40271-015-0154-8
Rate of colonoscopies with adenoma | With histology report, an average of 4 weeks after colonoscopy
  An adenoma was detected, resected and confirmed by the histology report in the colonoscopy.
Rate of colonoscopies with polyps | During colonoscopy
  Polyp detection in the colonoscopy as reported by the endoscopist.
Cecal intubation time | During colonoscopy
  Time expended in reaching the cecum
Withdrawal time | During colonoscopy
  Time expended in the withdrawal from cecum till the anus.
Information perceived quality assessed by a likert scale | The day of the colonoscopy just before beginning
  Perceived quality of the instructions and education received for the colonoscopy preparation by the participant. Assessed using a likert scale
Entry bowel cleansing as assessed by the modified Boston Bowel Preparation Scale | During colonoscopy (At the entry phase)
  Bowel cleansing during cecum intubation phase assessed using a modified Boston Bowel Preparation Scale which is without considering any additional cleansing during the endoscopy.
Rate of colonoscopies with flat polyps | During colonoscopy
  Flat polyp detection defined by Paris criteria: no polypoid nor ulcerated (Paris 0-IIa/b/c) in the colonoscopy as reported by the endoscopist.

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Machlab, Principal Investigator — Corporació Sanitaria Parc Taulí. Universidad Autónoma de Barcelona.
Locations (5):
- Spain (5):
  - Hospital de Mataró. Consorci Sanitari del Maresme., Mataró, Barcelona
  - Hospital Universitari Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Consorci Sanitari de Terrassa, Terrassa
  - Hospital Universitary Mutua de Terrassa, Terrassa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Machlab S, Martinez-Bauer E, Lopez P, Ruiz-Ramirez P, Gomez B, Gimeno-Garcia AZ, Pujals MDM, Tanco S, Sargatal L, Perez B, Justicia R, Enguita M, Pique N, Valero O, Calvet X, Campo R. Restrictive diets are unnecessary for colonoscopy: Non-inferiority randomized trial. Endosc Int Open. 2024 Mar 7;12(3):E352-E360. doi: 10.1055/a-2256-5356. eCollection 2024 Mar. PMID 38464979